CLINICAL TRIAL: NCT07175935
Title: A Prospective, Multicenter Registry Study of Amyotrophic Lateral Sclerosis in Thailand
Brief Title: Amyotrophic Lateral Sclerosis Registry in Thailand
Acronym: Thai ALS Regis
Status: Recruiting | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Jakkrit Amornvit, MD., Priciple Investigator, Chulalongkorn University
Other Study IDs: COA No. 0262/2025; NST (Other Grant/Funding Number: The Neurological Society of Thailand)
Record Dates: First submitted 2025-08-27; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: Amyotrophic Lateral Sclerosis; Epidemiological; Natural History
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational, multicenter registry designed to collect comprehensive clinical, genetic, and outcome data from patients diagnosed with amyotrophic lateral sclerosis (ALS) across Thailand. The registry will establish a national dataset to describe epidemiology, clinical presentation, progression, and treatment outcomes, and will serve as a platform for future clinical and translational research.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal neurodegenerative disorder that affects upper and lower motor neurons, leading to progressive muscle weakness, disability, and respiratory failure. Despite increasing research worldwide, Thailand lacks large-scale systematic data on ALS epidemiology, clinical characteristics, genetic profiles, and outcomes.

This registry will prospectively enroll ALS patients from major academic hospitals and specialized neuromuscular centers nationwide. Patients will be followed longitudinally using standardized assessments, including ALSFRS-R, staging systems (King, MiTos, 9-point), motor and respiratory function, quality-of-life measures, and cognitive/behavioral evaluations.

Data will be collected through a REDCap electronic database, ensuring confidentiality and compliance with Thai PDPA and international data protection standards. No experimental interventions will be performed; patients will receive standard of care treatments as determined by their treating physicians.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS according to El Escorial or Gold Coast criteria
* Age ≥ 18 years
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Patients unwilling to provide informed consent
* Patients with alternative diagnoses mimicking ALS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ALS patients attending university hospitals, tertiary neuromuscular clinics, and referral hospitals in Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 10 years
  Time Frame: From enrollment until death from any cause (assessed continuously, with updates at each follow-up).
  Outcome: Overall survival in ALS patients across Thailand, with survival curves stratified by demographic, clinical, and genetic factors.

SECONDARY OUTCOMES:
ALS Functional Decline | 10 years
  Measure: Change in ALS Functional Rating Scale-Revised (ALSFRS-R) score.
  Time Frame: Every 6-12 months.
  Outcome: Rate of functional decline, expressed as points lost per month/year.
Disease Staging Progression | 10 years
  Measure: King's and MiToS staging systems, 9-point staging.
  Time Frame: Every 6-12 months.
  Outcome: Proportion of patients progressing to higher stages; median time to stage transitions.
Respiratory Outcomes | 10 years
  Measure: Forced vital capacity (FVC % predicted).
  Time Frame: Every 6-12 months.
  Outcome: Decline in FVC
Changes in health-related quality of life over time. | 10 years
  Measure: EQ-5D-5L.
  Time Frame: Annually.
  Outcome: Changes in health-related quality of life over time.
Cognitive and Behavioral Profile | 10 years
  Measure: Edinburgh Cognitive and Behavioral ALS Screen (ECAS)
  Time Frame: Annually.
  Outcome: Frequency and pattern of cognitive/behavioral impairment in ALS patients.
Genetic and Environmental Risk Associations | 10 years
  Measure: Frequency of ALS-associated genetic variants (e.g., SOD1, C9orf72, TARDBP, FUS) and correlation with clinical phenotype and progression.
  Time Frame: As available.
  Outcome: Genotype-phenotype correlation; association with disease onset, progression, and survival.
Healthcare Utilization and Treatment Patterns | 10 years
  Measure: Use of riluzole, edaravone, non-invasive ventilation, gastrostomy, and multidisciplinary ALS clinic care.
  Time Frame: Throughout follow-up.
  Outcome: Patterns of treatment access and their association with survival and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial hospital, The Thai Red Cross Society, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results of this study (including clinical, demographic, and outcome measures) will be made available to qualified researchers upon reasonable request, following publication of the primary results. Access will be provided to investigators whose proposed use of the data has been approved by an independent review committee to ensure scientific merit and compliance with ethical standards. Data will be shared through secure data transfer under a data sharing agreement that protects participant confidentiality. Supporting documents, including the study protocol, statistical analysis plan, and informed consent form, will also be made available where applicable.
Supporting Information: Study Protocol, CSR
Time Frame: IPD will be available beginning 6-12 months after publication of the primary results and for up to 5 years thereafter.
Access Criteria: Requests for access should be directed to the Principal Investigator via institutional contact email. Applicants will be required to submit a research proposal outlining objectives, methods, and intended use of the data. Approval will be contingent on adherence to ethical and scientific standards, and execution of a data sharing agreement.